CLINICAL TRIAL: NCT05189600
Title: Can Waveform and Flow Traces From Mechanical Insuflattion:Exsufflation (MI:E) be Used to Identify Laryngeal Responses to MI:E and Thus Optimise Treatment Algorithms?
Acronym: SETTLE
Status: Recruiting | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Private Physiotherapy Education Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: 140484
Record Dates: First submitted 2021-09-14; First posted 2022-01-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Mechnical Insufflation:Exsufflation — Cough Augmentation device

SUMMARY:
Objectives:

* To establish if physiotherapists can use the waveform traces from the cough assist machine to work out when patients are having an abnormal airway response to cough assist
* To establish how cough assist device settings, particularly in breath and cough pressures affect a patient's response to using the cough assist device
* To provide some clinical guidance to physiotherapists on methods for assessing and treating abnormal airway responses to cough assist devices

Methodology:

Subjects will complete breathing tests; spirometry, peak cough flow (PCF) and sniff nasal inspiratory pressure (SNIP) to establish baseline breathing function and rule out anyone with breathing conditions. A nasal camera will be used to look at the voice box at rest.

Cough assist will be delivered via a face mask which will allow for simultaneous use of the nasal camera and cough assist carried out in the same way as another research team have done previously. The nasal camera will be attached to a video camera to allow recording, analysis and documentation of the observations. The cough assist protocol will be delivered by a physiotherapist experienced in delivering cough assist. Cough assist waveforms will be downloaded into Care Orchestrator software (Philips Respironics, Murraysville, USA) and reviewed at the same time as the nose camera recordings to establish if voice box responses can be identified from the waveform patterns. For confirmation of Care Orchestrator software waveforms, a device that records airflow during breathing (spirometer) will be connected (Alpha touch, Vitalograph, Ennis, Ireland) into the cough assist circuit in the same way another research team has before.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuromuscular disease(NMD) including but not limited to Motor Neurone Disease (MND), Multiple Sclerosis (MS) and Muscular Dystrophy
* Age ≥18

Exclusion Criteria:

* Unable to comply with protocol
* Unable to give informed consent
* Evidence of obstructive airways disease FEV1:FVC <0.7
* Patients with a history of:
* Un-drained pneumothorax
* Severe bronchospasm
* Head injury with ICP > 25mmHg
* Severe arterial hypotension
* Trache-oesophageal fistula
* Significant haemoptysis
* Facial fractures
* Vomiting
* Flail segment
* Epistaxis within two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuromuscular disease including but not limited to Motor Neurone Disease (MND), Multiple Sclerosis (MS) and Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
E70 (Mechnical insufflation:exsufflation) waveforms from Care Orchestrator | duration of study, approx. 30minutes per patient
  E70 (Mechnical insufflation:exsufflation) waveforms from Care Orchestrator
Nasal endoscopy video recordings. | duration of study, approx. 30minutes per patient
  Nasal endoscopy video recordings.waveforms.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansell SK, Parry R, Shah A, Gowing F, Greenfield C, Bhatt Y, Mandal S. Pilot observational cohort study to determine whether waveform and flow traces from mechanical insufflation-exsufflation (MI-E) can be used to identify laryngeal responses to MI-E and thus optimise treatment algorithms in neuromuscular patients in a tertiary centre: a protocol description. BMJ Open Respir Res. 2024 Mar 9;11(1):e001599. doi: 10.1136/bmjresp-2022-001599. PMID 38460974